CLINICAL TRIAL: NCT06996418
Title: Experimental Evaluation of Intergenerational Mealtime at a Shared Site: A Randomized Wait-listed Controlled Trial
Brief Title: Intergenerational Mealtime at a Shared Site: A Small-scale Trial
Acronym: IGM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Nestlé Nutrition Spain (Industry); Macrosad (Unknown)
Responsible Party: Principal Investigator, Mariano Sánchez, Head, Macrosad Chair in Intergenerational Studies, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 30C0647400
Record Dates: First submitted 2025-05-09; First posted 2025-05-30 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Healthy Nutrition; Intergenerational Relations; Well-being; Relational Care; Eating; Mealtimes
Keywords: Healthy Nutrition; Nutritional Knowledge; Intergenerational Mealtime; Intergenerational Shared Sites
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intergenerational Dining Room (Group #1) (Experimental): This is a group composed of 5 older people and 5 toddlers, all of them regular attendees at an intergenerational shared site.
  Interventions: Other: Intergenerational mealtime (intervention + follow-up)
- Intergenerational Dining Room (Group #2) (Experimental): This is a group consisting of 5 other older people and 5 toddlers (other than those in Intervention Group #1) from the same intergenerational shared site.
  Interventions: Other: Intergenerational mealtime (wait + intervention)
- Monogenerational Dining Room (Control Group) (No Intervention): This group is made up of 11 elderly people and 12 children from the same intergenerational shared site as the two intervention groups.

INTERVENTIONS:
Other: Intergenerational mealtime (intervention + follow-up) — Intergenerational lunchtime at an intentional intergenerational dining room 4 days a week for 8 weeks. Once this period is over, this group will move on to a follow-up phase that will last for another 8 weeks, during which they will eat 5 days a week in different dining rooms with their generational peers, as they had been doing up to the time of the intervention. Finally, they will undergo a last follow-up period of about 2 weeks.
  Arms: Intergenerational Dining Room (Group #1)
Other: Intergenerational mealtime (wait + intervention) — Waiting period consisting of 8 weeks (while Intervention Group #1 is using the intergenerational dining room). During this period toddlers and older people will eat lunch 5 days a week with their generational peers in separate dining rooms as they have been doing before the intervention. They will then move to eating together lunch 4 days a week for 8 weeks in the intergenerational dining room. Once this period is over they will enter a final follow-up phase for about 2 weeks during which they will go back to eat in generationally separate dining rooms.
  Arms: Intergenerational Dining Room (Group #2)

SUMMARY:
The goal of this study is to find out whether having children and older people who attend an intergenerational center eating lunch together on a regular basis may be an improvement over continuing to eat lunch with their generational peers in separate dining rooms at the center.

Specifically, the study analyzes the functioning and potential impact of an intergenerational dining room in terms of healthy eating, nutrition, self-evaluation of health and well-being, relational care, nutritional knowledge, and intergenerational attitudes. For this purpose, it sets up, in an intergenerational center, a dining room attended by children aged 2-3 years and older people aged 75 years and older who had previously been taking their lunch in separate dining rooms at the center.

The main questions this study aims to answer are:

* Does eating lunch at the intergenerational dining room improve the intake of healthy foods by children and older people compared to eating at their usual separate dining rooms with their peers?
* Does this type of intergenerational dining room serve as a space for nutritional education of children and older people?
* Does the experience of eating together have a positive influence in terms of children's attitudes towards older people and vice versa?

DETAILED DESCRIPTION:
The term Intergenerational Dining Room (IGD) refers to the intentional and planned space that enables people from different generations to periodically share the experience of eating together in settings dedicated to delivering care and development services (e.g. residential centers, schools), community work, intergenerational practices, etc.

The conceptual framework behind IGD has been articulated through combining the following three key components:

* Relationship-Centered Care (RCC): scientific evidence suggests that older people's care should focus on promoting meaningful relationships, rather than approaching them solely from the individualistic perspective of care.
* A life-course perspective on food: the act of feeding is a social practice that cuts across the life course and contributes to the construction of intergenerational relationships. Previous studies have pointed to the importance of mealtime as a space for interaction and learning between generations.
* Commensality, education, and nutritional health in caregiving spaces: research has shown that intergenerational programs have the capacity to improve the nutrition of their participants and encourage healthy eating habits, especially in settings where access to adequate food may be a challenge.

However, despite the growing interest in these components, empirical evidence remains limited, especially for structured intergenerational mealtime interventions with rigorous evaluation of their impact. Hence the goal of this interventional study: to analyze and explain, for the case of a specific institutional context - lunchtime at an intentional shared site's intergenerational dining room - not only the type of food and nutrition patterns but also some of the processes, causal mechanisms, and impacts associated with the social act of eating lunch together as a routine intergenerational practice.

Participant population is integrated by toddlers (ages 2-3) and older people (ages 79 and above) who attend regularly a co-located Preschool and Adult Day Care Center at an intergenerational shared site.

Apart from the 3 main questions presented in the brief summary, the study shall pay attention to further questions as the following:

* Is the intergenerational dining room a space where relational care and social interactions are practiced more than at the usual separate dining rooms?
* Does the subjective perception of health and well-being improve in older people because of their participation in intergenerational meals compared to having lunch at their regular daycare dining room with generational peers?
* Do children show greater well-being and participation at lunchtime when they are at the intergenerational dining room compared to the school dining room?; 4) Overall, is the feeding experience at the intergenerational dining room more positive than at dining rooms where each generational group has lunch with generational peers?

Researchers will compare a group of toddlers and older adults having lunch together several days per week to a similar group eating lunch just with their peers to see if intergenerational mealtimes make any difference. It is expected that the total number of intergenerational meals over the 16 intervention weeks amounts to 60.

Design of this study corresponds to a randomized wait-listed controlled trial including two wait-listed intervention groups (due to limitation of space to accommodate more than 10 people at the intergenerational dining room) and one control group.

Participants in the intervention will:

* Intergenerational Dining Room - Group #1 (IG1): During 8 weeks, have lunch at the intergenerational dining room four times per week and once a week at the regular peer-based dining room. Then, move to the peer-based dining room to have lunch five days per week for another 8 weeks (follow-up period).
* Intergenerational Dining Room - Group #2 (IG2): Have lunch at the peer-based dining room five days per week for some 8 weeks (waiting period), then for the following 8 weeks eat lunch at the intergenerational dining room four times per week and once a week at the regular peer-based dining room.
* Monogenerational Dining Room - Control Group (CG): Have lunch at their regular peer-based dining rooms for 16 weeks.

Both the control and intervention groups will undergo a final follow-up period of around two weeks to determine the duration of the observed impacts.

ELIGIBILITY:
Inclusion Criteria (older people):

* Informed consent signed by each participant or his/her legal representative.
* Eating autonomy: Ability to feed oneself without continuous assistance from another person.
* Expected stay at the Intergenerational Center until July 2025.
* Negative certificate of Sexual Offenses (mandatory in case of contact with minors).
* Screening for nutritional risk, dysphagia and oral health: Exclusion of persons with severe untreated malnutrition, severe dysphagia or oral problems preventing chewing.
* Adequate cognitive status: mild or moderate cognitive impairment (rating ≤5 on the Global Deterioration Scale - GDS).

Inclusion Criteria (toddlers):

* Informed consent: Signature of the legal guardian authorizing participation in the study.
* Child's assent: Positive expression of willingness to participate.
* Feeding autonomy: Ability to eat without continuous assistance from an adult.
* Expected permanence in the Intergenerational Center until July 2025.

Exclusion Criteria (older adults):

* Advanced cognitive impairment (GDS > 5) affecting comprehension and social interaction.
* Severe dysphagia or oral health problems preventing normal feeding.
* Unstable medical conditions that limit intergenerational dining attendance.
* History of aggressive behavior or history of refusal to interact with children.
* Lack of consent or refusal to participate in any of the study assessments.

Exclusion Criteria (toddlers):

* Need for ongoing feeding assistance.
* Severe medical conditions affecting feeding or social participation (e.g. severe metabolic disease).
* Expectation of transfer or departure from the Intergenerational Center prior to completion of the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-07-07 (Estimated); Study Completion 2025-07-21 (Estimated)

PRIMARY OUTCOMES:
Intake of healthy foods by children and older people | Day-by-day change in leftovers from baseline to final follow-up (18 weeks)
  Application of the Comstock method for the assessment of leftovers through photographing each dish after ingestion and calculating the proportion of waste (0%, 25%, 50%, 75%, & 100%).
Nutritional education | Baseline, 8 weeks, 16 weeks and 18 weeks
  Ad hoc test for assessing nutritional knowledge (identification and classification of foods, and discrimination between frequently and sporadically consumed foods) using the Nutriplato®. A set of five nutritional education activities is used to test nutritional knowledge among older adults (as toddlers' tutors) and toddlers. The number of successes and failures in each activity is assessed at different times throughout the intervention period.
Toddlers' attitudes towards older people | Baseline, 8 weeks, 16 weeks and 18 weeks
  A Visual Analog Scale (Young Children's Views of Older People) with original illustrations depicting images of older people according to a set of 11 bipolar pairs of adjectives (e.g., slow-fast, dull-exciting) will be presented to toddlers for them to locate their current attitudes towards older people. For each pair of adjectives ranging from -25 (extremely negative) to +25 (extremely positive) a mean global score will be calculated. Higher scores will indicate more positive attitudes towards older people.
Older people's attitudes towards toddlers | Baseline, 8 weeks, 16 weeks and 18 weeks
  Semantic differential with 9 pairs of bipolar adjectives with Likert-type responses (4 options). For each pair of adjectives ranging from -4 (extremely negative) to +4 (extremely positive) a mean global score will be calculated. Higher scores will indicate more positive attitudes towards toddlers.
Older people's attitudes about intergenerational exchanges | Baseline, 8 weeks, 16 weeks and 18 weeks
  Intergenerational Exchanges Attitude Scale , including 13 statements in two subscales ("Attributes to children" and "Relationships between older adults and children" subscales), each rated by older people along a 4-point Likert scale. This format allocates points from 4 (completely agree) to 1 (completely disagree). Higher scores indicate a more positive attitude in relation to intergenerational exchanges.

SECONDARY OUTCOMES:
Reaction to food items | Daily from week 4 to week 16
  Due to the young age of toddlers participating in the study, and based on a validated protocol, a member of the team will record observations and feedback on toddlers' reactions, facial expressions, and comments about foods at the moment of consumption. This additional measure will help to better contextualize and interpret results from the Comstock method (see primary outcome measure 'Intake of healthy foods by children and older people').
Relationship-centered environment | 4 weeks, 8 weeks, 12 weeks and 16 weeks
  Three components [Social Interactions, Mealtime Relational-Care Checklist, and Mealtime Clean-up] from the Mealtime Scan+ instrument, a reliable tool, will lead to assess both the social environment of the dining room and how relationship-centred were meals being observed. An overall quality of dining environment rating on a 1-8 scale will be calculated too.
Subjective well-being (older people) | 4 weeks, 8 weeks, 12 weeks and 16 weeks
  The WHO-5 Well-being Inde is a self-report instrument measuring mental well-being. It consists of 5 statements rated on a 4-point scale. The higher the score, the greater the well-being. A score below 8 indicates low well-being.
Toddlers' prosocial behavior | Baseline, 8 weeks and 16 weeks
  Prosocial Behavior subscale from the "Measure of Early Childhood Empathy" completed by toddlers' parents and teacher. It consists of 9 statements rated on a 4-point scale. The higher the score, the greater the prosocial behavior.
Place-based eating experience (older adults) | 4 weeks, 8 weeks, 12 weeks, & 16 weeks
  Ad hoc semi-structured qualitative interviews to older adults covering themes such as relationality, care and feeding experience; attention and knowledge about feeding; physical and emotional well-being; generational intelligence and views on toddlers.
Self-esteem (older people) | 4 weeks, 8 weeks, 12 weeks, 16 weeks
  Adapted and validated version of the Rosenberg's Self-Esteem Scale for older people. It consists of 5 statements in which older people self-rate along a 4-point Likert scale. Higher scores indicate higher self-esteem.
Subjective health (older people) | 4 weeks, 8 weeks, 12 weeks, 16 weeks
  EQ-5D's visual analogue scale records the respondent's self-rated health on a vertical 0-100 scale whose endpoints are 'Best imaginable health state' and 'Worst imaginable health state'.
Place-based eating experience (toddlers) | 4 weeks, 8 weeks, 12 weeks, & 16 weeks
  Ad hoc dialogue-based qualitative interviews to toddlers in the intervention groups exploring feeding experience, physical and emotional well-being and views on older people.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Sánchez, Doc.Soc., Principal Investigator — Universidad de Granada
Locations (1):
- Centro Intergeneracional de Referencia de Macrosad, Albolote, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided
A decision on IPD sharing will be made at a later date. It is a matter still to be discussed by the project stakeholders.

REFERENCES:
- See also: Public presentation of the pilot's launching (Spanish) — https://catedras.ugr.es/macrosad/informacion/noticias/macrosad-nestle-ugr-comedores-intergeneracionales

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT06996418/Prot_SAP_ICF_000.pdf